CLINICAL TRIAL: NCT01958099
Title: Behavior Change by Families in a Pediatric Emergency Department After Receiving Injury Prevention Information From a Safety Specialist Compared to a Computerized Kiosk
Brief Title: Teaching Injury Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Ohio Department of Public Safety (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIN381904
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Injury Prevention
Keywords: Injury Prevention
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injury Prevention Specialist (Other)
  Interventions: Behavioral: Education
- Kiosk Intervention (Experimental)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education

SUMMARY:
The purpose of this project is to compare the costs, ability to effectively screen and distribute relevant safety information, and assess products purchased and behavior changed by families after meeting with an injury prevention specialist compared to using a computerized emergency department kiosk. There will be a significantly greater reported practice of safety behaviors by families who visit a pediatric emergency department after using a computerized kiosk for injury screening and providing tailored recommendations than when the prevention information is provided by an injury prevention specialist.

DETAILED DESCRIPTION:
In the past few years, physicians have been proposing that an emergency department visit may act as a "teachable moment" and emergency medicine physicians should educate families about injury prevention. With an epidemic number of injuries occurring, every health care provider should play some role in combating the problem. However, emergency departments can be busy and overcrowded, making it difficult for staff, in a cost efficient manner, to be able to provide families with the appropriate injury prevention information. Kiosks have been shown to be effective in a pediatric emergency department setting to determine the needs of families and to educate them about safety practices. Thus, computerized kiosks may offer a more cost effective alternative to educating families, compared to a staff member, about injury prevention in the emergency medicine setting and they would have the ability to reach more individuals during the non-high peak emergency department hours which are difficult to staff. Also, a computerized kiosk may be more effective in eliciting a behavior change than a staff person as families may be inclined to answer more freely when asked questions anonymously, allowing them to receive more detailed safety information. In addition, the kiosk provides direct recommendations about behavior changes based on parental responses in a very short time period. Typically, families only hear about a few behavior change recommendations when discussing with an injury prevention staff person in an emergency department setting due to time constraints and family interest. With more directed injury prevention information and detailed recommendations on behavior changes in a cost efficient manner, kiosks may prove to be more effective in having families practice safer behaviors after leaving the pediatric emergency department.

This is a comparative study performed in the emergency department of a level 1 pediatric trauma center during the normal business hours of the Safety Resource Center. Families entering the pediatric emergency department for care will be randomized on specific days of the week to receive IP information from an IP specialist or from a computerized kiosk in the waiting room. A twenty day block random numbers table will be used to determine which days families entering the ED will utilize the computerized kiosk and which days they will be screened by clinical research assistants (CRCs) and provided with safety instructions by an IP specialist.

ELIGIBILITY:
Inclusion Criteria:

* Any parent/legal guardian of a child between the ages of 0-14 presenting to the emergency department with an acuity level of 3, 4, or 5 (per CCHMC ED guidelines) as determined by a triage nurse will be eligible for participation.

Exclusion Criteria:

* Family with a child presenting to the emergency department with an acuity level of 1 or 2 as given by a triage nurse.
* Non-English speaking families
* A parent or legal guardian who is less than 18 years of age
* A parent or legal guardian with a child who is greater than 14 years old.
* Primary parent or guardian not present with the child being seen in the Emergency Department.
* Families who are unable or unwilling to complete follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change to Practice Safer Behaviors | 16 months
  To determine if families cared for in a pediatric emergency department will report practicing safer behaviors after their visit if provided with targeted injury prevention information by a waiting room computerized kiosk in comparison with an injury prevention specialist.

SECONDARY OUTCOMES:
Change in Use of Safety Equipment | 16 months
  To determine if families screened using a computerized kiosk in a pediatric ED will admit to purchasing and using safety equipment more often if provided with recommendations using a computerized kiosk compared to an injury prevention specialist.
Time Spent on Intervention | 16 months
  To compare the time spent to be screened and provided targeted safety recommendations from a computerized kiosk in a pediatric ED compared to an IP specialist in the same setting.
Patient Satisfaction | 16 months
  To look at patient satisfaction about the IP information received from a computerized kiosk in a pediatric ED versus an injury prevention specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Gittelman, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Gittelman MA, Pomerantz WJ, McClanahan N, Damon A, Ho M. A computerized kiosk to teach injury prevention: is it as effective as human interaction? J Trauma Acute Care Surg. 2014 Sep;77(3 Suppl 1):S2-7. doi: 10.1097/TA.0000000000000317. PMID 25153050